CLINICAL TRIAL: NCT00479102
Title: Effectiveness of Iron Supplementation in the Second Year of Life for Prevention of Iron Deficiency
Brief Title: Prevention of Iron Deficiency in 2nd Year of Life
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: sor448707ctil
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2007-05-25 (Estimated); Status verified 2007-05

CONDITIONS: Iron Deficiency; Anemia
Keywords: Iron supplementation; Babies; Prevention
MeSH Terms: conditions — Iron Deficiencies; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ferripel-3 - iron polysaccharide complex for prevention

SUMMARY:
Healthy babies(age 8-18 months) following a routine blood count, with no anemia or iron deficiency, will be randomly placed in two groups. Group 1 will receive a 3 months preventive dose of an iron preparation (Ferripel 3 iron polysaccharide complex). Group 2 will be followed up as a control group. Following a nutritional questionnair, parents of all babies will receive instruction regarding appropriate nutrition in the 2nd year of life. A follow-up blood count will be taken from all participating babies 3 months after recruitment. The study aims to evaluate effectiveness of iron supplementation in the 2nd year of life. The hypothesis is that babies who receive iron supplementation in the 2nd year of life are less likely to develop iron deficiency or anemia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy babies without iron deficiency

Exclusion Criteria:

* Babies with iron deficiency or chronic diseases, premature babies and babies with hereditary hematological disease

Ages: 8 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Shalev, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Clalit Health Services Child Health Center, Rahat, Israel